CLINICAL TRIAL: NCT03300232
Title: Adapting an Effective CBT for Comorbidity to a Computer-Delivered Format
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSYCH-2018-26640
Record Dates: First submitted 2017-08-03; First posted 2017-10-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder; Social Anxiety; Alcohol Use Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder; Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer-based VC-CBT (Experimental): Computer-based VC-CBT: Three, one-hour computerized therapy sessions delivered on an interactive computerized platform with therapy blocks dedicated to each of three primary modules/goals: 1) psycho-education, 2) skills learning, and 3) individualized practice
  Interventions: Behavioral: Computer-based VC-CBT

INTERVENTIONS:
Behavioral: Computer-based VC-CBT — Computer-based VC-CBT: Three, one-hour computerized therapy sessions delivered on an interactive computerized platform with therapy blocks dedicated to each of three primary modules/goals: 1) psycho-education, 2) skills learning, and 3) individualized practice

SUMMARY:
Up to one-half of those in treatment for alcohol use disorder (AUD) has a co-occurring anxiety disorder ("comorbidity"), a condition that marks a high degree of treatment resistance, severity and relapse risk in AUD treatment patients. The investigators conceptualize comorbidity as a feed-forward system ("vicious cycle", [VC]) of interacting negative affect/stress, drinking motives/behavior, coping skills deficits, environmental circumstances, and neurobiological adaptations. Based on this model, the investigators developed and validated the VC cognitive-behavioral therapy (VC-CBT) to disrupt this system at several key linkage points. In a recently completed randomized controlled trial (RCT), the investigators found that adding the VC-CBT to standard AUD inpatient treatment resulted in better alcohol outcomes 4 months following treatment than did adding an anxiety treatment or standard AUD treatment alone. With a number needed to treat (NNT) index of 8 (relative to standard AUD treatment alone), the VC-CBT could, if broadly disseminated, have a large positive impact on AUD treatment. Unfortunately, several significant barriers related to the resource- and expertise-intensive delivery of the VC-CBT limit its dissemination potential and, hence, the impact of this otherwise effective treatment. Therefore, to maximize the public health and scientific potential of the investigators work, the investigators propose to adapt the therapist-delivered VC-CBT to a computer-delivered format to facilitate reliable and economical dissemination of the VC-CBT while maintaining its established efficacy.

DETAILED DESCRIPTION:
The first phase of the work (Year 1) will be to adapt the 6-session therapist-delivered VC-CBT for delivery on an internet-based computer platform. This work will be done using a standard iterative process for developing e-content in partnership with local technology experts experienced in producing engaging and effective e-learning products. Approximately 5 patients will be employed in this phase. The second phase (Years 2 and 3) will be devoted to a single arm pilot trial to test the efficacy of the refined computer-delivered VC-CBT. The investigators will recruit AUD treatment patients with co-occurring anxiety disorder to receive the computer-delivered VC-CBT (50 patients). Participants will complete follow-up assessments one and four months following treatment. Participants will rate user satisfaction and will be evaluated on skill and knowledge acquisition as well as use of the tools in the follow-up period. Success in the proposed work will serve as pilot data in support of a rigorous randomized clinical trial. The proposed work aims to provide an easy and inexpensive computer-delivered version of the VC-CBT that has comparable efficacy to the validated but resource-intensive therapist-delivered version. Achieving this will enable the VC-CBT therapy to benefit more AUD treatment patients and to be more easily studied by other investigators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-IV diagnosis of panic disorder (with or without agoraphobia), generalized anxiety disorder, or social anxiety disorder within the past 30 days
* Diagnostic and Statistical Manual-IV diagnosis of alcohol dependence within the last 30 days
* inpatient treatment at Lodging Plus primarily for alcohol (vs. other drug) dependence
* alcohol use in the 30 days preceding the beginning of their Lodging Plus (LP) treatment
* willingness and ability to provide informed consent
* minimum of a sixth grade English reading level (deemed necessary to complete study materials); as determined by their being able to read and understand the consent form
* familiarity with computer keyboarding as determined by history
* lives within reasonable driving distance of the Twin Cities and ability to travel to Fairview to allow for in-person follow-up interviews

Exclusion Criteria:

* Active psychosis or mania in the three months preceding the study
* Physical impairment (e.g., blindness, deafness) that interferes with study participation based on self-report or as judged by PI or study physician
* current significant suicide risk (i.e., intention and plan) as deemed by the PI and study physician to be serious and ongoing
* primary PTSD as determined by the Structured Clinical Interview for DSM (SCID) interview
* suspected cognitive impairment that interferes with study participation as informed by the SCID interview or as judged by the PI or study physician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
User ratings | up to 4 days post-treatment
  Likert scale ratings of understanding, engagement, and applicability to current problems
Knowledge Acquisition | up to 4 days post-treatment
  Multiple choice and True/False questions to assess knowledge communicated in program
Skills Acquisition | up to 4 days post-treatment
  Skill demonstration rated by study staff for accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Matt Kushner, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States